CLINICAL TRIAL: NCT04393025
Title: Endovascular Stenting of Medically Refractory Intracranial Arterial Stenotic (ICAS) Disease (Clinical and Sonographic Study)
Brief Title: Endovascular Stenting of Medically Refractory ICASD (Clinical and Sonographic Study)
Acronym: VasIntervent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Shafik Abdallah, Clinical professor of Neurology-Faculty of Medicine-ASU, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 142/2016
Record Dates: First submitted 2019-12-16; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Intervention Model Description: Two armed medical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intracranial Stenting (Other): 25 Patients presented with recurrent Ischemic CVS with Large ICSD received ICS
  Interventions: Device: Intracranial Stenting by Intracranial Stent Device
- Aspirin+Clopidogrel (Active Comparator): 25 Patients presented with recurrent Ischemic CVS with Large ICSD received optimal medical treatment
  Interventions: Drug: Optimum medical treatment

INTERVENTIONS:
Device: Intracranial Stenting by Intracranial Stent Device — Large Intracranial Vessels with ICSD underwent catheter lab and IC stent is inserted
  Other Names: cardiac and wingspan IC stent device
  Arms: Intracranial Stenting
Drug: Optimum medical treatment — Optimum Medical treatment
  Other Names: Clopidogrel 75 mg +Aspirin 161 mg
  Arms: Aspirin+Clopidogrel

SUMMARY:
Cerebral Endovascular Stenting of medically refractory Intracranial Stenotic Blood Vessels with Recurrent Ischemic Strokes patients

DETAILED DESCRIPTION:
Fifty patients were enrolled with 25 underwent Intracranial Stenting 25 received optimal medicall treatment without stenting and comparative study of primary outcome was conducted

ELIGIBILITY:
Inclusion Criteria:

1. Patients age between 30-80 years.
2. Symptomatic ICAS: presented with TIA or stroke, attributed to 70%-99% stenosis of a major intracranial artery: Internal carotid artery (ICA), middle cerebral artery (MCA) [M1segment], vertebral artery (VA), or basilar artery (BA).
3. Patient with recurrent TIA or stroke despite medical therapy, including anti-coagulation or antiplatelet and control of all vascular risk factors (DM, HTN and Hyperlipidemia).

Exclusion Criteria:

1. Patients previously stented at the target lesion or had extracranial stenosis.
2. Patient with acute stroke (within two weeks from the onset).
3. Complete occlusion of the artery on the imaging assessment.
4. Massive cerebral infarction (more than half the MCA territory), intracranial hemorrhage, epidural or subdural hemorrhage, and intracranial brain tumor on CT or MRI scans.
5. Contraindications to antithrombotic and/or anticoagulant therapies.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of IC stented patients in comparison to medically treated | 3 months
  clinical assessment by National Institute of Health Stroke Scale (NIHSS) for clinical impr
Functional improvement of IC stented patients in comparison to medically treated | 3 months
  Functional assessment by modified Rankin Scale (mRS) for functional improvement
Blood flow velocity accrossed Stenotic Large IC Vessels in comparison to medically treated | 3 months
  Transcranial doppler (TCD) assessment of Mean Flow Velocity (MFV) across IC vessels

SECONDARY OUTCOMES:
No Recurrent Ischemic stroke in stented ICSD patients | 6 months
  Clinical Assessment